CLINICAL TRIAL: NCT02264067
Title: Phase I Clinical Study of WAL2014 (Talsaclidine) Capsule: A Single Oral Dose Study
Brief Title: Pharmacokinetics and Safety of WAL2014 (Talsaclidine) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 506.111
Record Dates: First submitted 2014-10-13; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — talsaclidine fumarate

ARMS (2):
- Talsaclidine (Experimental): single rising doses
  Interventions: Drug: Talsaclidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talsaclidine
  Arms: Talsaclidine
Drug: Placebo
  Arms: Placebo

SUMMARY:
To assess the pharmacokinetics and safety of WAL2014 capsules administered orally as a single dose to healthy adult male volunteers in double blind manner.

ELIGIBILITY:
Inclusion Criteria:

Subjects for the study are healthy male adult volunteers who meet all the inclusion criteria listed below and do not fall into the exclusion criteria.

1. Age: 20-30 years old
2. Body weight: 50-80 kg
3. Obesity index: within +/-20% of the standard body weight
4. Those who have received screening examinations listed in protocol within one month prior to the start of the clinical study and have been judged as eligible by the investigator. Results of the simple test for gastric acidity are not used as the basis of the judgment.
5. Those who belong to volunteer members' association which has an office in Clinical Pharmacology Center, Ohsaki Clinic

Exclusion Criteria:

1. Those who have a history of allergic reaction or hypersensitivity to drugs
2. Those who have received any kind of drug(s) within one month prior to the administration of the investigational product
3. Those who have ingested alcoholic drink within two days before the administration of the investigational product
4. Those who have been admitted to a hospital, undergone surgery or donated blood within 3 months before the administration of the investigational product
5. Those who have participated in a phase I clinical study of a drug which contains a new active ingredient or a similar study within 4 months before the administration of the investigational product
6. Those who have a history of liver or renal disease
7. Those who are judged as ineligible for the clinical study by the investigator.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 1998-07; Primary Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) | up to 24 hours after drug administration
Time to reach maximum plasma concentration (tmax) | up to 24 hours after drug administration
Area under the plasma concentration-time curve (AUC) | up to 24 hours after drug administration
Distribution volume | up to 24 hours after drug administration
Total clearance | up to 24 hours after drug administration
Mean residence time (MRT) | up to 24 hours after drug administration
Urinary excretion rate | up to 24 hours after drug administration
Number of subjects with adverse events | up to 8 days after administration